CLINICAL TRIAL: NCT06456736
Title: Clinical Features and Prognostic Markers in Adult Patients With AE Requiring ICU Treatment
Status: Not yet recruiting | Type: Observational
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Lixia Qin, Principal Investigator, Central South University
Other Study IDs: Xiangya_critical AE
Record Dates: First submitted 2024-06-06; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Autoimmune Encephalitis
MeSH Terms: conditions — Autoimmune Diseases of the Nervous System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: None, non-interventional study — Not applicable, non-interventional study

SUMMARY:
Autoimmune encephalitis (AE) is a potentially life-threatening inflammation of the central nervous system (CNS) and constitutes 20%-30% of encephalitis cases in adults AE often leads to subacute, severe, and debilitating encephalitis necessitating long-term management in a neurologic intensive care unit (ICU). This study aims to explore the predictive factors for poor clinical outcomes by analyzing the clinical characteristics and prognosis of adult patients with critical AE requiring ICU admission. Prospective observational single center study in neurologic ICU, the second Xiangya hospital, Central South University. All patients admitted to the ICU for probable or confirmed AE (2022 Chinese guidelines for diagnosis and treatment of AE) will be included. Factors associated with a poor prognosis will be identified by multivariate analysis using a logistic regression.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as either ''definite'' or ''probable'' AE based on Chinese guidelines for diagnosis and treatment of AE (version 2022)
* Age ≥ 15 years
* Admission to an adult ICU during the course of the disease

Exclusion Criteria:

* Missing data on primary outcome
* ICU length of stay of 24 hours or less.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 200 patients admitted to the ICU for AE.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale | 12 months
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. It has become the most widely used clinic. mRS is scored on a scale of 0 to 6. The higher the score, the worse the prognosis

SECONDARY OUTCOMES:
Mortality | 12 months
  Rate of death at 12 months
Rate of complications | 12 months
  Septic shock, hyponatremia

IPD SHARING:
Plan to Share IPD: No